CLINICAL TRIAL: NCT00393497
Title: A Pilot Study of VEGF Inhibition in Patients With Lymphedema Following Breast Cancer Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0606-24; IUCRO-0162
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Breast Cancer; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab — Bevacizumab 15 mg/kg IV every 21 days

SUMMARY:
The purpose of this study is to evaluate the effectiveness of bevacizumab in women with lymphedema as a result of previous treatment for breast cancer.

DETAILED DESCRIPTION:
The primary objective of this study is:

• To assess the degree of improvement in arm edema as measured by changes in arm volume in patients with ipsilateral lymphedema

The secondary objectives of this study are:

* To assess the degree of improvement in arm edema as measured by changes in arm interstitial fluid pressure (IFP)
* To assess the degree of improvement in arm edema as measured by changes in extracellular fluid (ECF) volume based on bioelectrical impedance analysis (BIA) by lymphometer
* To assess the safety and tolerability of VEGF inhibition in this patient population
* To assess the clinical benefit in patients with ipsilateral lymphedema treated with vascular endothelial growth factor (VEGF) inhibition by evaluating patient responses to a quality of life questionnaire (FACT-B+4 lymphedema questions)
* To determine the impact of VEGF inhibition on circulating VEGF levels in patients with lymphedema

ELIGIBILITY:
Inclusion Criteria:

1. Have unilateral lymphedema of the ipsilateral arm attributed to prior surgical treatment or radiation therapy for breast cancer that is severe enough to warrant therapy in the opinion of the subject and treating physician.
2. All subjects must have greater than a 3 cm total difference in arm circumference between the affected and unaffected arm measured at five defined points:

   * each hand just distal to the thumb
   * each wrist at its narrowest point
   * each arm 30 cm proximal to the tip of the middle finger
   * each arm 40 cm proximal to the tip of the middle finger
   * each arm 50 cm proximal to the tip of the middle finger (if possible before the axilla is reached.)
3. Be at least 18 years of age
4. Have adequate organ function as specified below:

   * AST and ALT less than or equal to 2.0 times ULN
   * Total bilirubin less than or equal to 1.5 mg/dL
   * Serum creatinine less than or equal to 1.5 mg/dL
   * Urine protein:creatinine ratio < 1.0*
   * LVEF > institutional limits of normal by MUGA or ECHO
   * PT INR < 1.5; PTT < 1.5 x normal
   * Absolute neutrophil count greater than or equal to 1000/mm3
   * Platelets greater than or equal to 100,000/mm3
5. Agree to use effective contraceptive methods during the course of the study if the subject has child-producing potential
6. Have an ECOG performance status of 0 or 1

Exclusion Criteria:

1. Subjects must not be pregnant, lactating, or refuse to use appropriate birth control
2. Subjects must not have an active infection requiring parenteral or oral antibiotics
3. Subjects must not have clinically significant cardiovascular or cerebrovascular disease, including:

   Any history of:
   * Cerebrovascular disease including TIA, stroke or subarachnoid hemorrhage
   * Ischemic bowel
   * Hypertensive crisis or hypertensive encephalopathy Within the last 12 months
   * Myocardial infarction
   * Unstable angina
   * New York Heart Association (NYHA) grade II or greater congestive heart failure
   * Grade II or greater peripheral vascular disease
   * DVT or PE Active at study entry
   * Uncontrolled hypertension defined as SBP > 150 or DBP > 100
   * Uncontrolled or clinically significant arrhythmia.
4. Subjects may not have locally recurrent or metastatic disease
5. Subjects may not require concurrent therapeutic anticoagulation. (NOTE: Prophylactic doses of coumadin to maintain patency of a vascular access device is allowed). In addition, subjects with a bleeding diathesis are excluded.
6. Subjects may not have had major surgery within 4 weeks of starting protocol therapy (NOTE: Placement of a vascular access device is not considered major surgery)
7. Subjects may not have received radiation therapy, chemotherapy or trastuzumab within the past 6 weeks (NOTE: Concurrent adjuvant hormonal therapy is allowed.)
8. Subjects may not have altered the physical therapy regimen for lymphedema within the past month
9. Subjects may not have an indwelling venous device in the ipsilateral arm
10. Subjects may not have bilateral lymphedema
11. Subjects may not have a non-healing wound, ulcer or bone fracture.
12. Subjects may not have a known hypersensitivity to any component of Bevacizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Arm Volume | baseline, Day 1, Day 22, q 6wks, termination
The affected and unaffected arm measured at five defined points: | baseline, Day 1, Day 22, q 6wks, termination
each hand just distal to the thumb | baseline, Day 1, Day 22, q 6wks, termination
each wrist at its narrowest point | baseline, Day 1, Day 22, q 6wks, termination
each arm 30 cm proximal to the tip of the middle finger | baseline, Day 1, Day 22, q 6wks, termination
each arm 40 cm proximal to the tip of the middle finger | baseline, Day 1, Day 22, q 6wks, termination
each arm 50 cm proximal to the tip of the middle finger (if possible before the axilla is reached.) | baseline, Day 1, Day 22, q 6wks, termination
The volume of each arm will be calculated from these measurements using the Casley Smith method29. Treatment will be considered efficacious if there is a greater than or equal to 25% decrease in excess arm volume (affected arm volume minus unaffected arm | baseline, Day 1, Day 22, q 6wks, termination
Patients will initially be treated for 42 days (6 weeks). | Day 1-42

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States